CLINICAL TRIAL: NCT01569282
Title: Double Bypass vs Stent Strategy in Peroperatively Diagnosed Irresectable Pancreatic Cancer - A Prospective Randomized Multicenter Study
Brief Title: Double Bypass Versus Stent-treatment in Irresectable Pancreatic Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties to recruit patients
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Double bypass vs Stent
Record Dates: First submitted 2012-03-16; First posted 2012-04-03 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Pancreatic Cancer; Periampullary Tumor
Keywords: Surgical bypass; Hepaticojejunostomy; Gastrojejunostomy; Biliary stent; Enteral stent
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gastroenterostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Double bypass (Active Comparator)
  Interventions: Procedure: Hepaticojejunostomy and gastroenterostomy
- Stent Strategy (Active Comparator)
  Interventions: Procedure: Stent strategy

INTERVENTIONS:
Procedure: Hepaticojejunostomy and gastroenterostomy — Standard surgical techniques
  Other Names: Biliodigestive anastomosis; Gastrojenunal anastomosis
  Arms: Double bypass
Procedure: Stent strategy — Biliary and/or enteral stents on demand
  Other Names: Bile duct stent; Gastroduodenal stent; Enteral stent
  Arms: Stent Strategy

SUMMARY:
Double bypass (hepaticojejunostomy + gastrojejunostomy) is compared to stent strategy in patients planned for curative pancreatic resection in whom peroperative findings makes resection impossible.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperatively

   * Patients with stent treated tumor in the pancreatic head or periampullary planned for pancreaticoduodenectomy
   * The patient jaundice should have worn off and there should be no signs of duodenal obstruction
   * The patient has given informed consent after verbal and written information in accordance with approved ethics application
   * The patient has no anatomical conditions making endoscopic therapy impossible such as previous Billroth II or Gastric Bypass.
2. Intraoperatively

   * Peroperative findings of of carcinomatosis, metastases or local irresectability who oppose radical surgery
   * Surgical double bypass should be technically feasible
   * The patient has given informed consent after verbal and written information in accordance with approved ethics application

Exclusion Criteria:

* Peroperative signs of dysfunction on biliary stent
* Peroperative findings of gastric outlet obstruction
* Surgical double bypass not technically feasible

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2015-04-30 (Estimated); Study Completion 2015-10-31 (Estimated)

PRIMARY OUTCOMES:
Morbidity | Day 1-30 after randomization
  Initial morbidity in association to the laparotomy using the Clavien-Dindo Classification.

SECONDARY OUTCOMES:
Quality of life | Preop, 1 month postop and every third month
  Using the EORTC:s QLQ-C30 and QLQ-PAN26 questionaries
Numbers of readmissions to hospital | Up to two years after the laparotomy
The numbers of Surgical, Radiological or Endoscopical therapeutic re-interventions | Up to 24 months after the randomization
  The numbers of surgical, radiological or endoscopical interventions due to jaundice or gastric outlet obstruction from date of randomization until the date of death from any cause, whichever came first, assessed up to 24 months"

CONTACTS AND LOCATIONS:
Overall Officials: Lars Fändriks, Professor, Study Chair — Göteborg University; Claes Jönsson, Ass. Prof., Principal Investigator — Gothenburg Universitity
Locations (6):
- Sweden (6):
  - Department of Surgery, Sahlgrenska University Hospital, Gothenburg
  - Department of surgery, University Hospital, Linköping
  - Department of Surgery, Skane University Hospital, Lund
  - Department of Surgery, University Hospital, Örebro
  - Gastro Center Surgery, Karolinska University Hospital, Stockholm
  - Department of Surgery, University Hospital, Umeå